CLINICAL TRIAL: NCT02067702
Title: Effects of Limb Cooling on Essential Tremor.
Brief Title: Limb Cooling in Essential Tremor
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201300662
Record Dates: First submitted 2014-02-14; First posted 2014-02-20 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Limb Cooling Assessment of ET Control: Healthy, volunteers with no known dermatological lesions, sensitivity to cold, or peripheral vascular disease.
  Interventions: Procedure: Limb Cooling Assessment of ET
- Limb Cooling Assessment of ET Experimental: Patients with known essential tremor for at least a year, and +2 or worse action or kinetic tremor of one or both upper limbs involving at least the forearm and/or hand.
  Interventions: Procedure: Limb Cooling Assessment of ET

INTERVENTIONS:
Procedure: Limb Cooling Assessment of ET — The non-pharmacological treatment assessments of limb cooling will take place for the subjects which will include the upper limbs. Both clinical and physiological recordings will be measured for a difference in tremors at three different temperatures. 1)baseline assessment maintaining a normal body temperature (96-98°F). 2) at a temperature of 59°F and 3) at a temperature of 80°F for a period of 10 minutes. The clinical assessments will include the Tremor Rating Scale (TRS), Handwriting Assessment Battery (HAB) and the Functional Dexterity Test (FDT). In addition, the Bagnoli and Trigno EMG systems to record surface EMG signals from muscles and accelerometer readings.

SUMMARY:
Essential Tremor (ET) is characterized by tremors affecting the arms. The investigators will examine the effects of non-pharmacological limb cooling on clinical and physiological characteristics in patients presenting with ET at three different temperatures; and will measure changes in tremor amplitude after cooling of the upper limb.

DETAILED DESCRIPTION:
Once the subject has agreed to participate in the study the following assessments will be performed.

Three non-pharmacological assessments will be performed at different temperature to the upper limbs. The first will be a baseline assessment with upper limbs maintaining a normal body temperature (96-98°F). The second assessment will be performed with upper limbs at a temperature of 59°F and the third will be performed at a temperature of 80°F for a period of 10 minutes. At the end of 10 minutes, tremor measurements will be 15, 40, and 60 minutes.

1. Assessments will include the Tremor Rating Scale (TRS), Handwriting Assessment Battery (HAB) and the Functional Dexterity Test (FDT).
2. The Bagnoli and Trigno EMG systems will record surface EMG signals from muscles and accelerometer readings.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18 to 95 years,
* Clinical diagnosis of essential tremor for at least a year,
* A +2 or worse action or kinetic tremor of one or both upper limbs involving at least the forearm and/or hand

Exclusion Criteria:

* Dermatologic lesions in upper limbs (e.g. skin cancer, eczema, fresh or healing wounds, abrasions, acne, pustules, abscesses, or skin rash),
* Sensory loss in the upper limbs,
* Known history of sensitivity to cold (i.e., cold urticaria),
* Known peripheral vascular disease,
* Raynaud's phenomenon,
* Scleroderma

Healthy normal controls will be enrolled through advertisements. All controls will be examined to ensure that they are neurologically healthy.

The exclusion criteria for controls will remain same as those for patient subjects.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will enroll 24 subjects diagnosed with Essential Tremor (ET) and 24 subjects with no diagnosed of ET.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2014-10; Primary Completion 2016-08 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Hand writing assessment battery on limb cooling at 60 minutes post-cooling | 60 minutes post-cooling.
  Handwriting assessment battery includes pen control and manipulation subtests showed high to perfect agreement (line drawing subtest, κ = 1.0; dot subtest, κ = 0.80). The speed subtest showed perfect agreement (ICC = 1.0). Writing legibility showed high agreement for all five subtests (ICC = 0.71-0.83).
Tremor rating scale on limb cooling at 40 minutes post-cooling | 40 minutes post-cooling.
  Tremor Rating Scale (TRS), consists of 11 items that evaluate tremor in the head, arms, and legs. The rater assigns a score of 0 to 4 for each item, in ascending order of severity.
Functional dexterity test on limb cooling at 60 minutes post-cooling | 60 minutes post-cooling.
  Functional Dexterity Test (FDT) two scores are obtained: (1) time, in seconds, to complete the test and (2) combined total time with penalty seconds added to the initial time. If the patient exceeds 55 seconds, he or she receives a non-functional rating.
Hand writing assessment battery on limb cooling at 15 minutes post-cooling | 15 minutes post-cooling.
  Handwriting assessment battery includes pen control and manipulation subtests showed high to perfect agreement (line drawing subtest, κ = 1.0; dot subtest, κ = 0.80). The speed subtest showed perfect agreement (ICC = 1.0). Writing legibility showed high agreement for all five subtests (ICC = 0.71-0.83).
Hand writing assessment battery on limb cooling at 40 minutes post-cooling | 40 minutes post-cooling.
  Handwriting assessment battery includes pen control and manipulation subtests showed high to perfect agreement (line drawing subtest, κ = 1.0; dot subtest, κ = 0.80). The speed subtest showed perfect agreement (ICC = 1.0). Writing legibility showed high agreement for all five subtests (ICC = 0.71-0.83).
Tremor rating scale on limb cooling at 15 minutes post-cooling | 15 minutes post-cooling.
  Tremor Rating Scale (TRS), consists of 11 items that evaluate tremor in the head, arms, and legs. The rater assigns a score of 0 to 4 for each item, in ascending order of severity.
Functional dexterity test on limb cooling at 15 minutes post-cooling | 15 minutes post-cooling.
  Functional Dexterity Test (FDT) two scores are obtained: (1) time, in seconds, to complete the test and (2) combined total time with penalty seconds added to the initial time. If the patient exceeds 55 seconds, he or she receives a non-functional rating.
Functional dexterity test on limb cooling at 40 minutes post-cooling | 40 minutes post-cooling.
  Functional Dexterity Test (FDT) two scores are obtained: (1) time, in seconds, to complete the test and (2) combined total time with penalty seconds added to the initial time. If the patient exceeds 55 seconds, he or she receives a non-functional rating.
Tremor rating scale on limb cooling at 60 minutes post-cooling | 60 minutes post-cooling.
  Tremor Rating Scale (TRS), consists of 11 items that evaluate tremor in the head, arms, and legs. The rater assigns a score of 0 to 4 for each item, in ascending order of severity.

SECONDARY OUTCOMES:
Effect of limb cooling on the physiological characteristics of essential tremors. | 60 minutes post-cooling.
  To determine the physiological change in response to limb cooling, secondary outcome measures will include surface electromyography (EMG) with accelerometry.
Effect of limb cooling on the physiological characteristics of essential tremors. | 40 minutes post-cooling.
  To determine the physiological change in response to limb cooling, secondary outcome measures will include surface electromyography (EMG) with accelerometry.
Effect of limb cooling on the physiological characteristics of essential tremors. | 15 minutes post-cooling.
  To determine the physiological change in response to limb cooling, secondary outcome measures will include surface electromyography (EMG) with accelerometry.

CONTACTS AND LOCATIONS:
Overall Officials: Aparna W Shukla, M.D, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Movement Disorders Center, Gainesville, Florida, United States

REFERENCES:
- See also: Related Info — http://movementdisorders.ufhealth.org/